CLINICAL TRIAL: NCT05003167
Title: Effectiveness of Expiratory Muscle Strength Training for Improving Communication in ALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, HuberLab, Professor, SLHS, Purdue University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2020-524; 1F31DC019281-01 (NIH)
Record Dates: First submitted 2021-07-06; First posted 2021-08-12 (Actual); Results first posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: All participants enrolled will receive the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Expiratory Muscle Strength Training (Experimental): All participants will forcefully breathe out into an Expiratory Muscle Strength Training device (EMST-150) 25 times per day for 6 weeks. The EMST device will be set at a moderate intensity level (50% of each participant's maximum expiratory pressure).
  Interventions: Device: Expiratory Muscle Strength Training (EMST-150)

INTERVENTIONS:
Device: Expiratory Muscle Strength Training (EMST-150) — All participants will forcefully breathe out into an Expiratory Muscle Strength Training device (EMST-150) 25 times per day for 6 weeks. The EMST device will be set at a moderate intensity level (50% of each participant's maximum expiratory pressure).

SUMMARY:
A tele-health treatment study for individuals with early stage ALS with the aim to improve communication, cough response, and respiratory strength. All participants complete a respiratory strength training program using an Expiratory Muscle Strength Training (EMST 150) device from the comfort of their homes for 6 weeks.

DETAILED DESCRIPTION:
The investigators are looking for people with early stage ALS to participate in a completely tele-health (no in-person visits required) treatment study examining the effects of an Expiratory Muscle Strength Training device (EMST-150) on communication, cough, and respiratory strength. Participants will be required to attend 2 virtual baseline assessment sessions followed by 12 additional virtual training sessions (2 per week for 6 weeks). Participants should plan to be actively enrolled in the study for ~10 weeks (3 weeks of baseline monitoring followed by 6 weeks of training). Participants will also be required to fill out a series of questionnaires assessing the EMST's effectiveness via tele-health.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ALS
* Within the early stages of disease progression (i.e., able to talk, breathe, and eat independently)
* Speaker of English
* Have a family member/caregiver willing to assist as needed
* Have access to an electronic device and internet for tele-health

Exclusion Criteria:

* A history of neurological disease (besides ALS)
* A history of asthma or respiratory problems (e.g., COPD, emphysema)
* A history of head, neck, or chest surgery (except mastectomy)
* A history of smoking within the last 5 years
* Reliance on mechanical ventilation (including CPAP)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica E Huber, Ph.D., Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Expiratory Muscle Strength Training
Started | 13
Completed | 12
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Expiratory Muscle Strength Training
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.46 (8.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13
ALSFRS-R baseline [Mean (Standard Deviation); unit: units on a scale] — Amyotrophic Lateral Sclerosis Function Rating Scale-Revised (ALSFRS-R) (Cedarbaum et al., 1999) was used to assess overall physical functionality related to ALS. The survey requires participants to rate how 12 physical functions are impacted by their ALS (speech, salvation, swallowing, handwriting, etc). Participants are provided with a 4-point Likert scale to rate whether they still have complete control of that function (4) or no ability to perform that function (0). Total scores range from 0 to 48, with lower scores indicating more severe symptoms and higher scores and less severe symptoms.
  units on a scale | 38.8 (3.75)
Montreal Cognitive Assessment baseline [Mean (Standard Deviation); unit: units on a scale] — Montreal Cognitive Assessment 4.1 (MoCA) (Nasreddine et al., 2005) was used to screen cognition for inclusion. Scores range from 0-30. Scores over 25 are considered to reflect cognition that is within normal limits.
  units on a scale | 28.23 (1.42)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Post-treatment for Maximum Expiratory Pressure
Description: Change in expiratory muscle strength throughout the study duration measured by the participant blowing into a pressure meter
Time Frame: Baseline 2 (week 2), Pre-Training (week 3), and Post-Training (week 10)
Population: All participants with baseline, pre-training, and post-treatment maximum expiratory pressure values were included. The second baseline and pre-training values were averaged to obtain the pre-training value which was used along with the week 10 value (post-treatment).
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Expiratory Muscle Strength Training
Number analyzed (Participants) | 12
cmH2O
  Pre-training average | 66.10 (41.77)
  Post-training (week 10) | 83.75 (45.99)
Statistical Analysis 1: Comparison: Expiratory Muscle Strength Training; A mixed model ANOVA with session (pre-post-training) as a main effect and participant as a random factor was run via SAS 9.4. Alpha was set at .05; Test type: Superiority; p = .001, ANOVA; F = 8.48

2. Secondary Outcome: Peak Expiratory Flow Rate
Description: Change in cough strength (as measured by peak expiratory flow rate) throughout the study duration, measured using a flow meter that the participant coughs into - single coughs. Data from baseline 2 and pre-training were averaged for the pre--training value.
Time Frame: Baseline 2 (week 2), Pre-training (week 3), Post-Training (week 10)
Population: All participants with baseline 2 (week 2) and pre-training values (week 3) and post-training (week 10) data were included.
Measure: Mean (Standard Deviation); unit: liters per minute
Arm/Group | Expiratory Muscle Strength Training
Number analyzed (Participants) | 12
liters per minute
  Pre-training average | 265.97 (141.47)
  Post-training (week 10) | 273.47 (127.69)

3. Secondary Outcome: Change From Baseline to Post-Treatment in Utterance Length
Description: Change in utterance length (# of syllables produced on one breath) throughout the study duration. Participant read the Rainbow Passage and data were collected from this task.
Time Frame: Baseline 1 (week 1) and Post-Training (week 10)
Population: All participants who had baseline and post-training values for this measure. Data from the first baseline and the week 10 post-treatment value were used.
Measure: Mean (Standard Deviation); unit: syllables
Arm/Group | Expiratory Muscle Strength Training
Number analyzed (Participants) | 12
syllables
  Baseline (reading) - week 1 | 10.76 (3.29)
  Post-training (reading) - week 10 | 10.39 (4.11)
Statistical Analysis 1: Comparison: Expiratory Muscle Strength Training; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .113, ANOVA; df = 2,44; F = 2.29

4. Secondary Outcome: Change From Baseline to Post-Treatment in Number of Pauses
Description: Change in the total number of pauses that included breathing (breath pauses). Participant read the Rainbow Passage and data were collected from this task.
Time Frame: Baseline 1 (week 1) and Post-Training (week 10)
Population: All participants with baseline and post-training values. Data from the first baseline and the week 10 post-treatment value were used.
Measure: Mean (Standard Deviation); unit: number of pauses
Arm/Group | Expiratory Muscle Strength Training
Number analyzed (Participants) | 12
number of pauses
  Baseline (reading) - week 1 | 15.89 (8.28)
  Post-training (reading) - week 10 | 16.75 (10.99)
Statistical Analysis 1: Comparison: Expiratory Muscle Strength Training; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .052, ANOVA; F = 3.17

5. Secondary Outcome: Change From Baseline to Post-Treatment in Syntactic Location of Pauses
Description: Change in the location of pauses while breathing produced while reading. We determined where participants took breaths while reading the Rainbow Passage and categorized them according to syntax. Categories included at a major boundary (at the end of an independent clause marked by a period) and at a boundary that is not related to syntax (not a major or minor syntactical location). The number of pauses at each category of boundaries were converted to a percent of the total breaths taken while reading the passage.
Time Frame: Baseline 1 (week 1) and Post-Training (week 10)
Population: All participants with baseline and post-training values. Data from baseline (week 1) and post-training (week 10) were used.
Measure: Mean (Standard Deviation); unit: percent of pauses at the boundary
Arm/Group | Expiratory Muscle Strength Training
Number analyzed (Participants) | 12
percent of pauses at the boundary
  Baseline, major boundaries | 47.12 (37.59)
  Post-training, major boundaries | 46.09 (18.92)
  Baseline, boundaries unrelated to syntax | 8.71 (13.09)
  Post-training, boundaries unrelated to syntax | 12.33 (17.36)
Statistical Analysis 1: Comparison: Expiratory Muscle Strength Training; A mixed model ANOVA with session (pre-post-training) as a main effect and participant as a random factor was run via SAS 9.4. Alpha was set at .05. Results here are for percent of breaths at major boundaries; Test type: Superiority; p = .931, ANOVA; F = .07
Statistical Analysis 2: Comparison: Expiratory Muscle Strength Training; A mixed model ANOVA with session (pre-post-training) as a main effect and participant as a random factor was run via SAS 9.4. Alpha was set at .05. Results reflect percent of breaths at boundaries unrelated to syntax; Test type: Superiority; p = 0.164, ANOVA; F = 0.23

6. Secondary Outcome: Telehealth Satisfaction
Description: Participants rated 15 statements with a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). Example statements include: I can easily talk to my health-care provider, I can hear my health-care provider clearly, I can see my health-care provider as if we met in person, I think the care provided via telemedicine is consistent, and I receive adequate attention, telemedicine provides for my health care need, and overall, I am satisfied with the quality of service being provided via telemedicine. Total scores range from 0-75 and individual statement scores ranged from 1-5, with higher scores indicating higher satisfaction with the telepractice modality.
Time Frame: Post-Training (week 10)
Population: Only assessed at post-training. Included all participants who completed the scale. Higher values reflect more satisfaction and the score maximum is 75.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Expiratory Muscle Strength Training
Number analyzed (Participants) | 12
score on a scale | 60.58 (7.69)

7. Secondary Outcome: Change From Pre-Training to Post-Training in Communication Participation Item Bank
Description: Participants were instructed to use a 4-point Likert scale (3: not at all; 2: a little; 1: quite a bit; 0: very much) to rate if/how their ALS impacts ten hypothetical communicative situations. Participants total scores were then added together, ranging from 0-30, and converted to a T-score ranging from 24.2-71.0. High scores are more favorable, indicating that the participant feels that ALS impacts their communicative participation less than those with lower scores.
Time Frame: Pre-Training (week 3) and Post-Training (week 10)
Population: All participants with pre- and post-training scores. Data from the pre-training in week 3 and the week 10 post-treatment value were used.
Measure: Mean (Standard Deviation); unit: T-score scale points
Arm/Group | Expiratory Muscle Strength Training
Number analyzed (Participants) | 12
T-score scale points
  pre-training (week 3) | 47.78 (15.96)
  post-training (week 10) | 48.51 (14.65)

8. Secondary Outcome: Change From Baseline to Post-Treatment in ALS Quality of Life Scale
Description: The ALS Quality of Life Scale-Revised (ALSQOL-R) (Simmons, 2015) was used to measure how ALS impacts their quality of life in six domains: negative emotion, interaction with people and the environment, intimacy, religiosity, physical symptoms, and bulbar function. Participants rate whether they strongly disagree (0) or strongly agree (10) with 46 statements. Each domain score is given an average value between 0 (worse) and 10 (best). Total scores on the ALSQOL-R range from 0-460, but an average score ranging from 0-10 is computed by dividing the total score by the total number of items completed by the participant (usually 46). Higher scores reflect a higher quality of life. A survey assessing how each participant feels ALS impacts quality of life, and how that changes throughout the study duration. Total scores range from 0-460, with higher scores indicating greater contributions of ALS to quality of life.
Time Frame: Baseline 1 (week 1) and Post-Training (week 10)
Population: All participants with pre- and post-training scores on the scale. Lower scores reflect less effect of ALS on quality of life.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Expiratory Muscle Strength Training
Number analyzed (Participants) | 12
units on a scale
  pre-training | 5.97 (0.99)
  post-training | 5.94 (0.94)

9. Secondary Outcome: ALS Function Rating Scale Revised
Description: A survey that quantifies change in disease progression throughout the study duration. Participants rate how 12 physical functions are impacted by their ALS. For each function, participants are provided with a 4-point Likert scale to rate whether they still have complete control of that function (4) or no ability to perform that function (0). Total scores range from 0 to 48, with lower scores indicating more severe symptoms and higher scores and less severe symptoms.
Time Frame: Baseline 1 (week 1) and Post-Training (week 10)
Population: All participants with baseline (week 1) and post-training (week 10) scores were included.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Expiratory Muscle Strength Training
Number analyzed (Participants) | 12
score on a scale
  Baseline (week 1) | 39 [36 to 47]
  Post-training (week 10) | 37 [30 to 47]

10. Secondary Outcome: Psychosocial Impact of Assistive Devices Scale
Description: A survey assessing how the training device/modality impacts patient's psychosocial functions. The PIADS includes 12 items for competence, 6 for adaptability, and 8 for self-esteem. Participants use a 7-point Likert scale to rate the impact of a device on each item: a maximum negative impact (-3), somewhat negative impact (-2 or -1), zero impact (0), somewhat positive impact (1 or 2), maximum positive impact (3). Total scores range from -78 (maximum negative impact) to 78 (maximum positive impact).
Time Frame: Post-treatment (week 10)
Population: All participants with a post-treatment (week 10) score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Expiratory Muscle Strength Training
Number analyzed (Participants) | 12
score on a scale | 28.08 (26.61)

11. Secondary Outcome: Tele-health Session Attendance
Description: % of training sessions scheduled and attended by participants throughout the study duration
Time Frame: Measured at the end of training across the entire training period
Population: Participants who completed the training protocol
Measure: Mean (Standard Deviation); unit: percentage of sessions attended
Arm/Group | Expiratory Muscle Strength Training
Number analyzed (Participants) | 12
percentage of sessions attended | 95.37 (7.43)

12. Secondary Outcome: Adherence to Training Protocol
Description: Number of of training exhalations completed (25 exhalations into the device, 5 days per week) by participants throughout the study duration
Time Frame: Measured each week of training across the entire training duration
Measure: Mean (Standard Deviation); unit: percent of at-home training completed
Arm/Group | Expiratory Muscle Strength Training
Number analyzed (Participants) | 12
percent of at-home training completed | 90.65 (16.94)

ADVERSE EVENTS:
Time Frame: Over the course of the study (10 weeks for each participant)
Description: No changes to definitions of adverse events. Participants rated breathlessness on a scale of 0-10 (no breathlessness to completed breathlessness) before and after estimating maximum expiratory pressure and the EMST training protocol. Participants were also interviewed weekly about issues with at home training and were observed in training once a week.
Arm/Group | Expiratory Muscle Strength Training
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

LIMITATIONS AND CAVEATS:
The sample size was small. Participants enrolled in the current study likely had a preference or at least approval of telepractice prior to enrollment, since the recruitment materials stated that it was a telepractice study, and participants reached out to the researchers to express interest knowing that the study would be conducted through telepractice. Along similar lines, participants in the current study were highly educated and likely technologically savvy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT05003167/Prot_SAP_ICF_000.pdf